CLINICAL TRIAL: NCT02927522
Title: Donepezil Attenuate Postoperative Cognitive Dysfunction in Aged Patients- A Multi-center, Case Control, Randomized Clinical Trail
Brief Title: Donepezil Attenuate Postoperative Cognitive Dysfunction
Acronym: DAPOCD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Responsible Party: Principal Investigator, diansan su, Principal Investigator, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RJ20161003
Record Dates: First submitted 2016-10-05; First posted 2016-10-07 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis; Femoral Head Necrosis; Rheumatoid Arthritis
Keywords: Postoperative Cognitive Dysfunction; Donepezil; Hip replacement; Knee replacement; Postoperative delirium
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Postoperative Cognitive Complications; Emergence Delirium | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Placebo was administrated
  Interventions: Drug: Placebo
- Donepezil (Experimental): Donepezil (5mg/ day for 7 days) was administrated
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Donepezil a cholinesterase inhibitor, 5mg(1 pill)/ day for 7 days Po, was administrated from the day before surgery.
  Arms: Donepezil
Drug: Placebo — Placebo, 1 pill/ day for 7 days Po, was administrated from the day before surgery.
  Arms: Control

SUMMARY:
Postoperative cognitive dysfunction (POCD) occurs mainly in aged patients. POCD may increase the mortality and morbidity. However, the mechanism of POCD is not clear yet and no effective therapy method was proved. According to our previous study, the central cholinergic system impaired by the anesthesia and surgery play a very important role in the POCD and donepezil an acetylcholinesterase inhibitor can prevent the POCD after isoflurane anesthesia in aged mice. Donepezil is a commercial medicine used for the Alzheimer Disease, which is tolerable and has minimal adverse events. In present study a multi-center randomized case control study was conducted and we hypothesized that donepezil attenuate the POCD.

ELIGIBILITY:
Inclusion Criteria:

1. Elder than 60 years old
2. Speak Chinese Mandarin
3. Those who will undergo knee or hip replacement
4. Signed the inform consent
5. American Society of Anesthesiologists classification I to III

Exclusion Criteria:

1. Existing cerebral disease, or have a history of neurological and psychiatric diseases including Alzheimer Disease, stroke, epilepsy and psychosis;
2. existing cognitive impairment as evidenced by Mini-Mental State Examination scores below 24;
3. several audition or vision disorder;
4. unwillingness to comply with the protocol or procedures.
5. Can not communicated with Chinese Mandarin
6. Existing bradycardiac arrhythmia（Heart rate <60 bpm for any reasons）
7. Existing gastrointestinal ulcer
8. Existing urinary incontinence
9. Existing asthma or chronic obstructive pulmonary disease
10. Allegory to Donepezil

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of POCD 7 days(or before leaving hospital ) after surgery | 7 days after surgery or before leaving hospital
The incidence of postoperative delirium after surgery | 1 to 7 days after surgery

SECONDARY OUTCOMES:
POCD incidence 1 months after surgery | 1 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, M.D., Ph.D., Principal Investigator — RenJi Hospital
Locations (1):
- Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai, Shanghai Municipality, China